CLINICAL TRIAL: NCT01899898
Title: Phase 2/3 Study of a Simplified Modified Atkins Diet in Children With Refractory Epilepsy
Brief Title: Efficacy of a Simplified Modified Atkins Diet in Children With Refractory Epilepsy
Acronym: SMAD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Satinder Aneja, Director Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMAD
Record Dates: First submitted 2013-06-14; First posted 2013-07-16 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Refractory Epilepsy
Keywords: Refractory epilepsy; Dietary therapy; Non-Pharmacological therapy; Simplified Modified Atkins Diet
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Anticonvulsants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simplified Modified Atkins Diet (Experimental)
  Interventions: Other: Simplified Modified Atkins Diet
- Antiepileptic drugs alone (Active Comparator)
  Interventions: Drug: Antiepileptic drugs alone

INTERVENTIONS:
Other: Simplified Modified Atkins Diet — Modified Atkins diet with the following modifications:
  1. Pictorial representation of various food items and exchange lists will be provided.
  2. Instead of weights, we will provide standardized measures
  3. We will calculate the amount of carbohydrates of daily readily available foods in the standardized measures
  4. We will formulate recipes and diets based on locally available and culturally acceptable foods.
  5. We will develop a parent instruction manual.
  6. We will also develop methods for parents with low levels of literacy to maintain seizure logs. This will be done by using bars and color codes.
  7. We will develop methods for parents with low levels of literacy to measure and record urine ketones. This will be done by using color codes.
  Arms: Simplified Modified Atkins Diet
Drug: Antiepileptic drugs alone — The anti-epileptic drugs will be continued alone for 3 months following which they will be offered Simplified Modified Atkins Diet
  Arms: Antiepileptic drugs alone

SUMMARY:
One third of children with epilepsy have seizures that are medically intractable. Uncontrolled seizures pose a variety of risks to children, including higher rates of mortality, developmental delay and cognitive impairment. Epilepsy surgery is not a feasible option for most children with refractory epilepsy. The ketogenic diet and the modified Atkins diet have been shown to be effective alternative treatments in children with refractory epilepsy. However, these need parents to be educated, and understand complex instructions of weighing foods and diet preparation. Therefore, children with parents with low levels of literacy and poor socioeconomic status have not been able to benefit from these therapies. Also, the paucity of trained dieticians and limited availability of labeled foods in resource-constraint settings has made these dietary therapies even more inaccessible.

This study aimed to to develop a simple-to-administer variation of the modified Atkins diet for use in children with refractory epilepsy and to evaluate the efficacy and tolerability of this simplified modified Atkins diet in children with refractory epilepsy in a randomized controlled open-label trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 2 - 14 years.
2. Seizures persisting daily or more than 7 per week despite the use of at least 2 anti-epileptic drugs in appropriate doses and levels (whenever available) in suitable to the syndrome and EEG findings.

Exclusion Criteria:

1. Known or suspected inborn error of metabolism:

   Patients with clinical suspicion of metabolic disorder as evidenced by 2 or more of the following- a history of parental consanguinity, prior affected siblings, unexplained vomiting, intermittent worsening of symptoms, recurrent episodes of lethargy, altered sensorium, or ataxia, hepatosplenomegaly on examination With or without 2 or more of the following biochemical abnormalities High blood ammonia (>80mmol/L), High arterial lactate (>2 mmol/L), metabolic acidosis (pH <7.2), hypoglycaemia (blood sugar <40 mg/dl), abnormal urinary aminoacidogram, presence of reducing sugars or ketones in urine, and positive results on urine neurometabolic screening tests.

   In such patients, blood tandem mass spectrometry or urine gas chromatography mass spectroscopy (GCMS) will be obtained to look for inborn error of metabolism.
2. Surgically remediable causes of epilepsy such as tumors, cortical dysplasias, mesial temporal lobe epilepsy etc with refractory focal epilepsy.

   We will perform MRI brain, and short term video-EEG in all patients with focal seizures to look for surgically remediable causes.
3. Motivational or psychosocial issues in the family which would preclude compliance
4. Systemic illness- chronic hepatic, renal or pulmonary disease

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The proportion patients who achieve > 50% seizure reduction from the baseline in the simplified modified Atkins diet plus anti-epileptic drug therapy group at 3 months in comparison to the anti-epileptic drug therapy alone group | 3 months

SECONDARY OUTCOMES:
Tolerability and the adverse effects of the simplified modified Atkins diet | 3 months
  Tolerability of the diet and any adverse events will be evaluated by means of parental interview at each visit. Parents will be questioned for the following symptoms - vomiting, lethargy, poor appetite, refusal to feed and constipation in particular. Any other parental concerns will also be noted. The proportion of patients with each symptom in both the groups will be evaluated.

OTHER OUTCOMES:
Proportion of patients withdrawing from the simplified modified Atkins diet plus antiepileptic drug treatment group during the study period | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Satinder Aneja, MD, Principal Investigator — Pediatric Neurology, Department of Pediatrics, Lady Hardinge Medical College and Associated Kalawati Saran Children's Hospital
Locations (1):
- Division of Pediatric Neurology, Department of Pediatrics, Lady Hardinge Medical College and Associated Kalawati Saran Children's Hospital, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Martin-McGill KJ, Bresnahan R, Levy RG, Cooper PN. Ketogenic diets for drug-resistant epilepsy. Cochrane Database Syst Rev. 2020 Jun 24;6(6):CD001903. doi: 10.1002/14651858.CD001903.pub5. PMID 32588435